CLINICAL TRIAL: NCT04605952
Title: Study to Find the Percentage of Cases Retaining COVID-19 IgG Antibodies 45-65 After They Have Tested Positive
Status: Completed | Type: Observational
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, Senior Consultant, Tata Main Hospital, Tata Main Hospital
Other Study IDs: 152473
Record Dates: First submitted 2020-10-23; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 IgG antibody positive between 28th June to 15th July 2020: As a serosurveillance measure, 3296 asymptomatic employees of an industrial workforce Jamshedpur (India) were tested for SARS-CoV-2 IgG antibodies specific for the spike subunit antigen by the ErbaLisa COVID-19, Erba Corporate Services (United Kingdom) between 28th June and 15th July 2020. All those who initially tested SARS-CoV-2 IgG antibody positive were retested at 45-65 days
  Interventions: Diagnostic Test: Repeat SARS-CoV-2 IgG antibodies at 45-65 days

INTERVENTIONS:
Diagnostic Test: Repeat SARS-CoV-2 IgG antibodies at 45-65 days — All cases who initially tested positive for SARS-CoV-2 IgG antibodies would undergo a repeat test at 45-65 days

SUMMARY:
As a serosurveillance measure asymptomatic employees of an industrial workforce Jamshedpur (India) were tested for COVID-19 IgG antibodies. Of the tested employees who were positive for COVID-19 IgG antibodies the study aimed to find the percentage of cases who retained their COVID-19 IgG antibodies 45-65 days after initially testing positive.

DETAILED DESCRIPTION:
As a serosurveillance measure, 3296 asymptomatic employees of an industrial workforce Jamshedpur (India) were tested for COVID-19 IgG antibodies specific for the spike subunit antigen by the ErbaLisa COVID-19, Erba Corporate Services (United Kingdom) between 28th June and 15th July 2020.

The cases who tested positive for COVID-19 IgG antibodies were repeat tested for the presence of COVID-19 IgG at 45-65 days after initially testing positive. This was done with the aim of finding out the percentage of cases retaining their IgG antibodies at 45-65 days of initially testing positive.

ELIGIBILITY:
Inclusion Criteria:

SARS-CoV-2 IgG antibody positive between 28th June and 15th July 2020

Exclusion Criteria:

SARS-CoV-2 IgG antibody negative between 28th June and 15th July 2020

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asymptomatic workforce
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of cases retaining SARS-CoV-2 IgG antibodies at 45-65 days | 45-65 days
  Percentage of cases retaining SARS-CoV-2 IgG antibodies at 45-65 days

CONTACTS AND LOCATIONS:
Overall Officials: DR.DEB S NAG, MD, Principal Investigator — Tata Main Hospital
Locations (1):
- Dr.Deb Sanjay Nag, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: No